CLINICAL TRIAL: NCT05724758
Title: Patient Reported Outcomes After Oncoplastic Breast Conserving Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Brust-Zentrum AG (Other)
Responsible Party: Sponsor
Other Study IDs: Patient reported outcome
Record Dates: First submitted 2023-01-04; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer in Situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ | interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Breast-conserving surgery — Following oncoplastic surgeries are performed at the Brust-Zentrum in Zurich:
  * Oncoplastic reconstruction with round-block technique
  * Oncoplastic reconstruction using J-Plastic
  * Oncoplastic reconstruction using V-Plastic
  * Oncoplastic reconstruction using Grisotti
  * Oncoplastic reconstruction using Batwing
  * Oncoplastic reconstruction using Mammareductionplasty (Wise Pattern, Vertical)
  * Oncoplastic perforator flap surgery

SUMMARY:
The goal of this study is to assess patient satisfaction after oncoplastic breast conserving surgery. With the help of a breast-questionnaire the patient satisfaction will be assessed before the surgery and 4 weeks, 6 months and 1 year after the operation. The main question it aims to answer are: Does breast conserving surgery improve quality of life.

type of study: cohort study, observational

OCBS = oncoplastic breast conserving surgery BCT = breast conserving therapy DCIS = ductal carcinoma in situ

participant population/health conditions

* Patients with newly diagnosed breast cancer, that can be treated breast conserving
* the participants have to be at least 18 years old

Participants will fill out a questionnaire pre surgery, 4 weeks, 6 months and 1 year after the surgery. The individual questionnaires will be compared.

DETAILED DESCRIPTION:
The management of breast cancer has undergone a significant shift over the last century. The advances in systemic therapy have not only improved the overall prognosis however also allowed for less radical surgery and more breast conservable efforts. The term oncoplastic breast conserving surgery was first coined in the early 90s where breast cancer surgery was performed while incorporating plastic surgical techniques. Therefore, this enabled the preservation of the natural breast shape with good aesthetic outcomes. Over the years oncoplastic breast conserving surgery has become widely accepted and adopted into routine clinical practice by most breast cancer surgeons. The oncological safety surrounding oncoplastic breast conserving surgery have been well established. Rates of positive surgical margins and re-excision rates have been shown to be similar to traditional lumpectomy operations. Complication rates are also comparable and oncoplastic breast conserving surgery does not result in delays in adjuvant treatments. However, many surgeons would concur that the most significant benefit of oncoplastic breast conserving surgery (OBCS) is patient satisfaction and the potential improvement in their quality of life.

Patient reported outcomes (PROMs) allow us to objectively assess patient satisfaction and the impact the intervention has had onto their lives. Incorporating PROMs into daily clinical practice would not only facilitate shared-decision making but also allow us to tailor clinical management to suit individual patient needs. This study however also aims to assess the patient reported outcome after breast surgery and in the follow up time (after radiotherapy, ...).

ELIGIBILITY:
Inclusion Criteria:

* BCT oncoplastic surgery technique
* Women > 18 years

Exclusion Criteria:

* Previously treated ipsilateral breast cancer or DCIS
* Severe psychological illness by doctors' discretion (as taking part in a study could increase anxiety) or severe dementia, that stops them to consent to the procedure
* Pregnant women
* Distant metastatic disease (M1)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Brust-Zentrum Zürich undergoing oncoplastic breast surgery recruited between March and September 2023
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change of patient satisfaction with their breasts pre- and post breast-conserving surgery | before the surgery and 4 weeks after the surgery
  To assess patient satisfaction using BREAST-Q over the duration of the breast cancer clinical management and follow up i.e., pre-, and postoperative: 4 weeks, 6 months and 1 year after the surgery.
Change of quality of Life pre- and post breast-conserving surgery | before the surgery and 4 weeks after the surgery
  To assess Quality of Life using BREAST-Q over the duration of the breast cancer clinical management and follow up i.e., pre-, and postoperative: 4 weeks, 6 months and 1 year after the surgery.

SECONDARY OUTCOMES:
impact of age (>70 and < 60 years old) on Patient reported outcome measures | baseline and 4 weeks postoperative
  To assess the impact of age (> 70 and < 60 years old) on patient reported outcome measures (validated questionnaire) after oncoplastic surgery, If age has an impact on patient satisfaction with their breasts pre and post surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freites-Martinez A, Santana N, Arias-Santiago S, Viera A. Using the Common Terminology Criteria for Adverse Events (CTCAE - Version 5.0) to Evaluate the Severity of Adverse Events of Anticancer Therapies. Actas Dermosifiliogr (Engl Ed). 2021 Jan;112(1):90-92. doi: 10.1016/j.ad.2019.05.009. Epub 2020 Sep 3. No abstract available. English, Spanish. PMID 32891586
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Weigelt E, Scherb H. [Data protection and data access (I): federal data protection law and the social welfare code with reference to carrying out occupational medicine epidemiologic studies in Germany]. Gesundheitswesen. 1992 Nov;54(11):666-72. German. PMID 1286250
- [Background] McIntosh J, O'Donoghue JM. Therapeutic mammaplasty--a systematic review of the evidence. Eur J Surg Oncol. 2012 Mar;38(3):196-202. doi: 10.1016/j.ejso.2011.12.004. Epub 2011 Dec 27. PMID 22206704
- [Background] Carter SA, Lyons GR, Kuerer HM, Bassett RL Jr, Oates S, Thompson A, Caudle AS, Mittendorf EA, Bedrosian I, Lucci A, DeSnyder SM, Babiera G, Yi M, Baumann DP, Clemens MW, Garvey PB, Hunt KK, Hwang RF. Operative and Oncologic Outcomes in 9861 Patients with Operable Breast Cancer: Single-Institution Analysis of Breast Conservation with Oncoplastic Reconstruction. Ann Surg Oncol. 2016 Oct;23(10):3190-8. doi: 10.1245/s10434-016-5407-9. Epub 2016 Jul 12. PMID 27406093
- [Background] Rose M, Manjer J, Ringberg A, Svensson H. Surgical strategy, methods of reconstruction, surgical margins and postoperative complications in oncoplastic breast surgery. Eur J Plast Surg. 2014;37(4):205-214. doi: 10.1007/s00238-013-0922-4. Epub 2014 Feb 1. PMID 24659858
- [Background] Kaviani A, Sodagari N, Sheikhbahaei S, Eslami V, Hafezi-Nejad N, Safavi A, Noparast M, Fitoussi A. From radical mastectomy to breast-conserving therapy and oncoplastic breast surgery: a narrative review comparing oncological result, cosmetic outcome, quality of life, and health economy. ISRN Oncol. 2013 Sep 12;2013:742462. doi: 10.1155/2013/742462. PMID 24167743
- [Background] Wijgman DJ, Ten Wolde B, van Groesen NR, Keemers-Gels ME, van den Wildenberg FJ, Strobbe LJ. Short term safety of oncoplastic breast conserving surgery for larger tumors. Eur J Surg Oncol. 2017 Apr;43(4):665-671. doi: 10.1016/j.ejso.2016.11.021. Epub 2016 Dec 18. PMID 28041648
- [Background] Nizet JL, Maweja S, Lakosi F, Lifrange E, Scagnol I, Seidel L, Albert A, Jerusalem G. Oncological and surgical outcome after oncoplastic breast surgery. Acta Chir Belg. 2015 Jan-Feb;115:33-41. PMID 26021789
- [Background] Cil TD, Cordeiro E. Complications of Oncoplastic Breast Surgery Involving Soft Tissue Transfer Versus Breast-Conserving Surgery: An Analysis of the NSQIP Database. Ann Surg Oncol. 2016 Oct;23(10):3266-71. doi: 10.1245/s10434-016-5477-8. Epub 2016 Aug 12. PMID 27518043
- [Background] Klit A, Tvedskov TF, Kroman N, Elberg JJ, Ejlertsen B, Henriksen TF. Oncoplastic breast surgery does not delay the onset of adjuvant chemotherapy: a population-based study. Acta Oncol. 2017 May;56(5):719-723. doi: 10.1080/0284186X.2017.1281437. Epub 2017 Feb 6. PMID 28162018
- [Background] Rose M, Svensson H, Handler J, Hoyer U, Ringberg A, Manjer J. Patient-reported outcome after oncoplastic breast surgery compared with conventional breast-conserving surgery in breast cancer. Breast Cancer Res Treat. 2020 Feb;180(1):247-256. doi: 10.1007/s10549-020-05544-2. Epub 2020 Jan 27. PMID 31989380
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246
- [Background] Stolpner I, Heil J, Feisst M, Karsten MM, Weber WP, Blohmer JU, Forster T, Golatta M, Schutz F, Sohn C, Hennigs A. Clinical Validation of the BREAST-Q Breast-Conserving Therapy Module. Ann Surg Oncol. 2019 Sep;26(9):2759-2767. doi: 10.1245/s10434-019-07456-y. Epub 2019 May 21. PMID 31115853
- [Background] Cordova LZ, Hunter-Smith DJ, Rozen WM. Patient reported outcome measures (PROMs) following mastectomy with breast reconstruction or without reconstruction: a systematic review. Gland Surg. 2019 Aug;8(4):441-451. doi: 10.21037/gs.2019.07.02. PMID 31538070
- [Background] Lagendijk M, van Egdom LSE, van Veen FEE, Vos EL, Mureau MAM, van Leeuwen N, Hazelzet JA, Lingsma HF, Koppert LB. Patient-Reported Outcome Measures May Add Value in Breast Cancer Surgery. Ann Surg Oncol. 2018 Nov;25(12):3563-3571. doi: 10.1245/s10434-018-6729-6. Epub 2018 Sep 3. PMID 30178391
- [Background] Mundy LR, Homa K, Klassen AF, Pusic AL, Kerrigan CL. Breast Cancer and Reconstruction: Normative Data for Interpreting the BREAST-Q. Plast Reconstr Surg. 2017 May;139(5):1046e-1055e. doi: 10.1097/PRS.0000000000003241. PMID 28445351